CLINICAL TRIAL: NCT00534261
Title: Evaluation of the Correlation Between the MS Functional Composite Index and Two Quality of Life Scales (MS54 and AMS Quality of Life) in Relapsing MS Patients Treated With Interferon Beta-1a (AVONEX®)
Brief Title: Does Quality of Life Improve in Multiple Sclerosis Patients Treated With Interferon Beta-1a?
Acronym: FLAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIO-BNL 99-01
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2007-12-13 (Estimated); Status verified 2007-12

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Avonex; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): patients received Avonex IM injections and be evaluated for quality of life criteria
  Interventions: Drug: Interferon beta-1a

INTERVENTIONS:
Drug: Interferon beta-1a — IM injection

SUMMARY:
This study was to find out if patients with Relapsing Remitting Multiple Sclerosis treated with Interferon beta-1a had an improved quality of life after treatment with Interferon beta-1a

DETAILED DESCRIPTION:
The study was an open-label, multi-center, international post-marketing study (phase 4). Eligible patients were interferon naïve patients suffering from relapsing MS. The duration of a subject's participation in the study was up to a maximum 26 months.

ELIGIBILITY:
Inclusion Criteria:

* Relapsing Remitting Multiple Sclerosis
* Interferon naïve
* Eligible for interferon beta-1a (AVONEX®) therapy as per Summary of Product Characteristics:
* Subject has had relapsing MS for > 1 year
* Subject has had experienced 2 exacerbations in the last 2 years
* Subject had an EDSS [5] score of < 5.5
* Subject was ambulant

Exclusion Criteria:

* Diagnosis of MS defined as progressive
* History of any significant cardiac, hepatic, pulmonary, or renal disease; immune deficiency; or other medical conditions that would preclude therapy with interferon beta
* History of severe allergic or anaphylactic reactions or history of hypersensitivity to human albumin
* History of seizures within the 3 months prior to starting this study
* History of intolerance to acetaminophen (paracetamol), ibuprofen, naproxen or other NSAIDs, that would preclude use of at least one of these during the study
* History of intolerance to interferons
* Previous use of interferon beta
* Female subjects who were pregnant or breast-feeding
* For female subjects, unless postmenopausal or surgically sterile, unwillingness to practice effective contraception

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 1999-11; Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to evaluate the correlation between the MS Functional Composite Index and two Quality of Life scales (MS Quality of Life 54 and AMS Quality of Life) in patients treated with interferon beta-1a (AVONEX®). | screening, Day -30, Day -1, Months 3, 6, 12, 18, and 24

SECONDARY OUTCOMES:
Reproducibility of Quality of Life scales per language version | months 18 and 24
Reliability of the Quality of Life scales per language version | months 18 and 24
EDSS score throughout the study | screening, Day -1, Months 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Biogen-Idec Investigator, Principal Investigator — neurologyclinicaltrials@biogenidec.com
Locations (3):
- Coordinating Research Site, Sijsele-Damme, Belgium
- Coordinating Research Site, Esch-sur-Alzette, Luxembourg
- Coordinating Research Site, Glasgow, Scotland, United Kingdom